CLINICAL TRIAL: NCT06026904
Title: The Effects of Transcutaneous Auricular Vagus Nerve Stimulation on Motivation in Major Depressive Disorder With Anhedonia
Brief Title: The Effects of taVNS on Motivation in MDD With Anhedonia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Fengqiong Yu, Associate Professor, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Y&C
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: taVNS; anhedonia; intervention
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Intervention Model Description: This study will enroll two groups of patients with Major Depressive Disorder (MDD): one group will receive active transcutaneous auricular Vagus Nerve Stimulation (taVNS) treatment, while the other group will receive sham taVNS treatment (the same flow path, but targeting a different stimulation site).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Comparator: Real Stimulation (Active Comparator): The active Stimulation of taVNS lasted 30 mins. The stimulation protocol is preset to a biphasic impulse frequency of 25 Hz with a stimulation duration of 30 s, followed by a 30 s off phase. Behavior and ERPs datasets should be acquired before the first taVNS session and after the last taVNS session.The electrical current is transmitted by a titanium electrode placed at the cymba conchae.
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- Sham Comparator: Sham Stimulation (Sham Comparator): The active Stimulation of taVNS lasted 30 mins. The stimulation protocol is preset to a biphasic impulse frequency of 25 Hz with a stimulation duration of 30 s, followed by a 30 s off phase. Behavior and ERPs datasets should be acquired before the first taVNS session and after the last taVNS session.The electrical current is transmitted by a titanium electrode placed at the earlobe of the midpoint of the outer ear margin.
  Interventions: Device: transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — taVNS was developed as a non-invasive variant of VNS where the vagus nerve is stimulated through the skin of the auricle, which has become a promising avenue for research and, potentially, treatment of various disorders. Commonly, taVNS is applied via the ear targeting the auricular branch of the vagus nerve, where the stimulation elicits far-field potentials. In line with preclinical studies, acute taVNS enhances invigoration of effort and response inhibition capability.

SUMMARY:
Study of non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) intervention to improve the reward motivation and response inhibition of major depression disorder and its brain network mechanism.

DETAILED DESCRIPTION:
Anhedonia is the core symptom of MDD, which means they have deficits in processing rewards.MDD get lesser positive feelings than healthy controls from rewards as they could not use the reward outcome to update the value of a stimulus, which in consequence impedes their reward motivation or response inhibition and worsen their symptom. This study is dedicated to revealing how reward motivation or response inhibition ability could be intervened by taVNS intervention, which has been proven is highly relevant to reward motivation and response inhibition ability. Implementing a safer intervention of taVNS stimulation might help us to prove a better treatment for patients.

All patients underwent a medical evaluation that included physical examination and routine laboratory studies before and after taVNS stimulation treatment. Before and after the taVNS treatment, depression symptom of each participant was assessed by the Hamilton Depression Scale and the Beck Depression Self-Rating Scale. The anhedonia severity was evaluated by The Temporal Experience of Pleasure Scale, the Self-Report Apathy Evaluation Scale, the Positive Valence system scale and the Motivation and Pleasure Scale. The neuroimaging data are collected using event-related potentials during the effort reward task and stop signal task before and after the intervention. Patients were randomly allocated into an active group and a sham group. This study plans to enroll a minimum total sample size of 30 participants in active and sham group respectively according to the Power and Sample Size program. The decision to enroll a patient was always made prior to randomization. Each patient will be treated for 4 weeks with 25Hz taVNS. Each participant was interviewed in detail about the adverse event of the taVNS intervention during 10 days. Every participant should take part in the study voluntarily and sign an informed consent form before the study.

ELIGIBILITY:
Inclusion Criteria:

Meet the criteria of depression assessed by at least two psychiatrists according to the fifth version of Diagnostic and Statistical Manual of Mental Disorders.

The score of Hamilton Depression Rating Scale-17 is larger than 18 and the score of the Apathy Evaluation scale is lager than 37.

Patients were taking antidepressants--Selective Serotonin Reuptake Inhibitor(SSRIs) alone.

Age was between 18 to 60 year old. The education duration was at least 6 years.

The vision or corrected vision was normal.

Right handedness.

No treatment of rTMS, transcranial direct current stimulation, or electroconvulsive therapy before.

Exclusion Criteria:

History of significant head trauma or neurological disorders.

Alcohol or drug abuse.

Focal brain lesions.

History of seizure.

First degree relative with epilepsy, significant neurological illness or head trauma, endocrine disease.

Significant unstable medical condition.

Recent aggression or other forms of behavioral dyscontrol.

Left-handedness.

Pregnancy.

Current alcohol or drug abuse

Inability to provide informed consent.

Patients with contraindications or factors affecting imaging quality, such as pacemakers, cochlear implants, or hearts Cerebrovascular metal stent, and metal denture.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Scale | baseline;10days after treatment; 1month and 3 month post-treatment
  The participants' depression symptom assessed by the Hamilton Depression Scale change from baseline after the treatment. Score reference value: <7 points, no depression;7 to 17points, mild depression;18to 24 points, moderate depression; > 24 points, severe depression. If remission rate reaches 50%, the treatment will be considered effective.
Change from baseline in Apathy Evaluation Scale | baseline;10days after treatment; 1month and 3 month post-treatment
  The participants' reward motivation assessed by the Apathy Evaluation Scale change from baseline after the treatment. Score reference value: <37 points, no apathy; ≥37points, apathy. If remission rate reaches 25%, the treatment will be considered effective.

SECONDARY OUTCOMES:
The change from baseline in behavioral results of effort reward task | baseline;4 weeks post-treatment
  Behavioral results changed and discount parameters generated from the model change from baseline after the treatment.
The change from baseline in event-related brain potentials during the effort reward task | baseline;4 weeks post-treatment
  The amplitudes of brain potentials of reward-related positivity and P3 assessed by event-related brain potentials methods change from baseline after the treatment.
The change from baseline in behavioral results of stop signal task | baseline;4 weeks post-treatment
  Behavioral results changed from baseline after the treatment.
The change from baseline in event-related brain potentials during the stop signal task | baseline;4 weeks post-treatment
  Cue-evoked cue-P3 and N2 mean wave amplitude changes and latencies, as well as spectral intensities. Wave amplitude and latency of target-P3 and N2 evoked by target stimuli, and spectral activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, MD, Study Chair — Anhui Medical University; Fengqiong Yu, MD, Study Director — Anhui Medical University; Rong Ye, Phd, Study Director — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China